CLINICAL TRIAL: NCT04285099
Title: Frequency Effect of Subthalamic Nucleus Deep Brain Stimulation Through the Dual System on Freezing of Gait in Parkinson Disease
Brief Title: Frequency Effect of STN-DBS Through the Dual System on FOG in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H-1902-132-1091
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease, Freezing of Gait, Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Because our study is a double-blinded trial within one group, participant and investigator do not know whether the frequency is 130Hz or 60Hz.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients with FOG after STN-DBS[A] (Experimental): Initially started by A setting
  Interventions: Device: Application of dual system in frequency A
- PD patients with FOG after STN-DBS[B] (Experimental): Initially started by B setting
  Interventions: Device: Application of dual system in frequency B

INTERVENTIONS:
Device: Application of dual system in frequency A — The investigators set two values of frequency (130, 60Hz) in IPG and allow the patients to change the frequencies freely using the patient controller. Technician randomly sets 130 Hz, 60HZ to A or B.
  Arms: PD patients with FOG after STN-DBS[A]
Device: Application of dual system in frequency B — The investigators set two values of frequency (130, 60Hz) in IPG and allow the patients to change the frequencies freely using the patient controller. Technician randomly sets 130 Hz, 60HZ to A or B.
  Arms: PD patients with FOG after STN-DBS[B]

SUMMARY:
We aim to confirm the effect for FOG by changing the frequency through the dual-system approach in PD patients after STN-DBS.

DETAILED DESCRIPTION:
The investigators set two values of frequency (130, 60Hz) in IPG and allow the patients to change the frequencies freely using the patient controller. After four weeks, the investigators will check the UPDRS part I, II, IV, FOG-Q, and PDQ-39 values at each frequency, including the proportion of use of two frequencies.

ELIGIBILITY:
Inclusion Criteria:

* patients with PD who are aged 30 years or older
* patients with bilateral STN-DBS
* patients who have a FOG at their med "off" state in outpatient clinic or hospitalization, or UPDRS part II FOG subscore above 1

Exclusion Criteria:

* patients without FOG
* patients who have undergone DBS
* patients who have had previous brain surgery
* patients who have undergone reoperation of DBS
* patients who underwent unilateral DBS
* patients with cognitive impairment (MMSE <18)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Stimulation frequency ratio in 4 weeks | 4 weeks
  Proportion of two frequencies in 4 weeks

SECONDARY OUTCOMES:
Comparison of Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score in 130 and 60Hz at the fourth week | 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score will be used to compare 130Hz with 60Hz. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Comparison of Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score in 130 and 60Hz at the fourth week | 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score will be used to compare 130Hz with 60Hz. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Comparison of Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score in 130 and 60Hz at the fourth week | 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score will be used to compare 130Hz with 60Hz. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Comparison of Freezing of Gait Questionnaire score in 130 and 60Hz at the fourth week | 4 weeks
  Freezing of Gait Questionnaire score will be used to compare 130Hz with 60Hz. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Comparison of Parkinson's Disease Questionnaire-39 score in 130 and 60Hz at the fourth week | 4 weeks
  Parkinson's Disease Questionnaire-39 score will be used to compare 130Hz with 60Hz. Higher scores mean a worse outcome. [minimum 0, maximum 156]

CONTACTS AND LOCATIONS:
Locations (1):
- Beom S Jeon, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No